CLINICAL TRIAL: NCT05104099
Title: Evaluation of the Ability of PpIX Fluorescence to Mark High-grade Vulvar Intraepithelial Neoplasia Following the Methyl Aminolevulinate (Metvixia®) Application
Brief Title: Evaluation of New Diagnostic Tool Using Fluorescence to Detect High-grade Vulvar Intraepithelial Neoplasia
Acronym: PhotodiVIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-000568-31
Record Dates: First submitted 2021-09-29; First posted 2021-11-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-06

CONDITIONS: Vulvar Intraepithelial Neoplasia; Vulvar High Grade Squamous Intraepithelial Lesion; Differentiated Vulvar Intraepithelial Neoplasia
Keywords: Vulvar Intraepithelial Neoplasia; Vulvar High Grade Squamous Intraepithelial Lesion; Photodynamic diagnosis; Metvixia; Differentiated vulvar intraepithelial neoplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metvixia application for Photodynamic diagnosis (Experimental): Patients who benefit Metvixia application to the vulva to realize fluorescence guided biopsies (Photodynamic diagnosis).
  Interventions: Drug: Metvixia Topical Cream

INTERVENTIONS:
Drug: Metvixia Topical Cream — Metvixia is applied with a spatula, in a thick layer, to clinically visible lesions and all over the vulva. After applying the cream, the area will be covered with a bandage which should remain in place for 3 hours. After 3 hours of application, the bandage and the cream will be carefully removed. The application area will be cleaned and then immediately exposed to a continuous spectrum of light at a wavelength of 405 nm by a xenon lamp.
  The most fluorescent areas will be identified. Then in white light, the practitioner will perform at least two biopsies under non-topical local anesthesia in the area of application of Metvixia®: one in the fluorescent area and one in the non-fluorescent area.
  If there is no fluorescent labeling, two samples will be taken from two different non-fluorescent areas. In the event that all the zone is fluorescent , two samples will be taken from two different fluorescent zones.

SUMMARY:
This study is a single-center propsective clinical trial to assess the ability of fluorescence techniques to mark high-grade vulvar intraepithelial neoplasias including high-grade vulvar squamous intraepithelial lesions and differentiated vulvar intraepithelial neoplasias following 3 hours Metvixia application.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over,
* With isolated high-grade vulvar intraepithelial neoplasia OR associated with invasive cancer proven histologically by biopsy
* Naive of any vulvovaginal treatment (surgery or radiotherapy)
* No metastases
* WHO <or equal to 3
* Contraception method for women of childbearing potential
* Patient affiliated to the social security scheme
* Patient who understood, signed and dated the information note and the
* consent form,
* Patient able and willing to follow all study procedures in accordance with the protocol.

Exclusion Criteria:

* History of hypersensitivity to the active substance methyl aminolevulinate or to any of the components of the drug (including peanut oil and refined almond oil), soybean or peanut
* Ulceration or hyperpigmented lesions of the vulva
* Patient with porphyria
* Any previous vulvovaginal treatment (surgery or radiotherapy)
* Metastatic disease
* Patient undergoing treatment for any other invasive cancer
* Pregnant, likely to be or breastfeeding patient
* Patient deprived of liberty or under guardianship (including guardianship)
* Inability to undergo medical monitoring of the trial for geographic, social or psychological reasons.
* Patient already included in another therapeutic trial with an experimental molecule,
* Associated pathology that may prevent the patient from receiving METVIXIA application and light exposure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of the success of the photodynamic diagnosis | 14 days (+/- 4 days) after the photodiagnosis
  Percentage of patients for whom the procedure successfully demonstrated high-grade vulvar intraepithelial neoplasias in fluorescence confirmed by biopsy.
  A patient will be considered successful if the presence or absence of fluorescence is consistent with the anatomo-pathological result, that means if her sample in the fluorescent area is positive in pathology and her sample in the non-fluorescent area is negative in anatomo-pathology.
  For a patient with no fluorescent labeling, the pathological results of her two samples must be negative for the patient to be considered successful. For a patient where the entire area fluoresces, the anatomo-pathological result of her two samples must be positive for the patient to be considered successful.

SECONDARY OUTCOMES:
Sensitivity of the photodynamic diagnosis | 14 days (+/- 4 days) after the photodiagnosis
  The sensitivity will correspond to the number of fluorescent zones among the positive zones in anatomopathology.
Specifity of the photodynamic diagnosis | 14 days (+/- 4 days) after the photodiagnosis
  The specificity will correspond to the number of non-fluorescent zones among the negative zones in anatomo-pathology.
Intensity of flurescence evaluation | The day of the photo analysis with a specific software
  The fluorescence intensity will be measured by the signal to noise ratio, also called SNR (Signal to Noise Ratio) on photographie
Tolerance evaluation | At inclusion, after applying the cream for 3 hours, before and immediately after the blue light exposition and at and the final study visite (14 days +/- 4 after the photodiagnosis)
  The tolerance of the application will be assessed by the number of grade 3 to 5 toxicity. The toxicity will be evaluated using the CTCAE v5 scale (Common Terminology for Adverse Events). The different grade on this scale is 1 to 5 (1 correspond to a asymptomatic or mild symptome, 2 to moderate toxicity, 3 to severe or medically significant but not immediately life-threatening toxicity, 4 to life-threatening consequences or urgent intervention indicated and 5 to the death related to the toxicity.
Pain Evaluation | At inclusion, 1 hour after Metvixia application, before and immediately after the blue light exposition and at and the final study visite (14 days +/- 4 after the inclusion)
  Pain will be assessed using a numerical scale from 0 to 10 (0 corresponds to no pain and 10 to maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine HEJL, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No